CLINICAL TRIAL: NCT03570814
Title: Safety of the Co-administration of Azithromycin, Albendazole and Ivermectin Versus Standard Treatment Regimens During Mass Drug Administration (MDA) in Ethiopia: a Cluster-randomized Trial
Brief Title: Cluster RCT of Co-administration Azithromycin, Albendazole & Ivermectin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Armauer Hansen Research Institute, Ethiopia (Other); Federal Minstry of Health of Ethiopia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11985
Record Dates: First submitted 2018-06-04; First posted 2018-06-27 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-04

CONDITIONS: Trachoma; Lymphatic Filariases
MeSH Terms: conditions — Trachoma; Elephantiasis, Filarial

STUDY DESIGN:
Intervention Model Description: Cluster randomised trial. Approximately 40 clusters per study arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Separate Administration (Active Comparator): Standard administration of Albendazole/Ivermectin separated from administration of azithromycin
  Interventions: Drug: Administration of Albendazole on Day 1; Drug: Administration of Ivermectin on Day 1; Drug: Administration of Azithromycin on Day 15
- Co-administration (Experimental): Combined administration of Albendazole/Ivermectin/Azithromycin at a single time point
  Interventions: Drug: Administration of Albendazole on Day 1; Drug: Administration of Ivermectin on Day 1; Drug: Administration of Azithromycin on Day 1

INTERVENTIONS:
Drug: Administration of Albendazole on Day 1 — Participants will receive Albendazole 400mg on study day 1.
Drug: Administration of Ivermectin on Day 1 — Participants will receive Ivermectin 150mcg/kg (max 12mg) on study day 1. Doses of Ivermectin will be determined using a standard dosing pole.
Drug: Administration of Azithromycin on Day 1 — Participants will receive Azithromycin 20mg/kg (max 1gm) on study day 1. Doses of Azithromycin will be determined using a standard dosing pole.
  Arms: Co-administration
Drug: Administration of Azithromycin on Day 15 — Participants will receive Azithromycin 20mg/kg (max 1gm) on study day 15. Doses of Azithromycin will be determined using a standard dosing pole.
  Arms: Separate Administration

SUMMARY:
Cluster-randomised trial comparing co-administration of Azithromycin/Ivermectin/Albendazole with separate administration of Azithromycin and Ivermectin/Albendazole.

The study will be conducted in Beneshangul-Gumuz region, Ethiopia. Within this district, a study group of 8,000 people (in approximately 40 clusters) will receive the azithromycin, ivermectin & albendazole at a single time. A control group of 8,000 people (in approximately 40 clusters) within the same district will receive the current MDA treatment schedule beginning with Ivermectin/Albendazole followed two weeks later with azithromycin. All drug dosing will be in line with standard FMOH and WHO Guidelines for MDA for trachoma and lymphatic filariasis.

The study will randomly sort subdistrict communities (Gotes) into the trial arm and the control arm. The study will compare the number of adverse events (AEs) and severe adverse events (SAEs) between the two arms to determine if co-administration is not inferior to the standard treatment. The primary outcome will be to demonstrate the safety of the triple-drug administration as measured by incidence of AEs/SAEs following the MDA.

ELIGIBILITY:
Inclusion Criteria:

1. Residing in the community for at least three months;
2. Eligible to receive all three agents according to standard MDA criteria

Exclusion Criteria:

1. Not eligible to receive one or more drugs according to standard MDA criteria;
2. Less than 5 years of age (not eligible for ivermectin)**
3. Pregnant women (azithromycin only, not eligible for albendazole and ivermectin)
4. Lactating women (Only administered azithromycin and albendazole, not eligible for ivermectin)**
5. History of allergies to the drugs being studied (azithromycin, ivermectin, albendazole)
6. Residents who cannot swallow tablets

   * Note that patients that are not eligible for IVM, will receive azithromycin and albendazole. Patients that receive azithromycin and albendazole will be followed up through the same procedure as the triple drug therapy to try to track any AEs attributed to the two drug combination.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13511 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Self Reported Adverse Event | 1 Month
  The incidence of self-reported adverse events following MDA. We will collect data on the presence of common symptoms/signs prior to drug administration. All patients will be reviewed 24-48 hours after treatment and asked to report adverse events. We will calculate the proportion of newly occurring adverse events following treatment and calculate the whether the proportion of patients experiencing an adverse event differs between study arms,

SECONDARY OUTCOMES:
Cost of Administration Drug Separately compared to Cost of Co-Administration of Drugs | 1 month
  Analysis of the cost effectiveness of co-administration compared to separate administration of drugs
Community perceptions | 1 month
  An analysis of community perceptions of benefits of co-administration at a single time point vs standard separated MDA will be conducted by conducting focus groups and in-depth interviews with study participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Community Recruitment across whole district, Community Recruitment Across Whole District, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McPherson S, Tafese G, Tafese T, Behaksra SW, Solomon H, Oljira B, Miecha H, Debebe KA, Kebede B, Gebre T, Kebede F, Seife F, Tadesse F, Mammo B, Aseffa A, Solomon AW, Mabey DCW, Marks M, Gadisa E. Safety of integrated mass drug administration of azithromycin, albendazole and ivermectin versus standard treatment regimens: a cluster-randomised trial in Ethiopia. EClinicalMedicine. 2023 Apr 27;59:101984. doi: 10.1016/j.eclinm.2023.101984. eCollection 2023 May. PMID 37152362